CLINICAL TRIAL: NCT00134758
Title: Efficiency of Ursodesoxycholic Acid in the Treatment of Duodenal Adenomas in Familial Adenomatous Polyposis Patients. URSOPAF
Brief Title: Ursodeoxycholic Acid in the Treatment of Duodenal Adenomas in Familial Adenomatous Polyposis (FAP) Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Axcan Pharma (Industry)
Responsible Party: Christophe Aucan, Department of clinical research and development
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P030419; AOM 03041
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2009-07-29 (Estimated); Status verified 2009-07

CONDITIONS: Adenomatous Polyposis Coli, Familial
Keywords: Treatment of adenomas of the duodenum in FAP patients.; Adenoma
MeSH Terms: conditions — Adenomatous Polyposis Coli; Adenoma | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Ursodeoxycholic acid during 2 years :
  * between 40 and 50 kg : 500 mg/day
  * between 51 and 75 kg : 750 mg/day
  * between 76 and 100 kg : 1000 mg/day
  Interventions: Drug: Ursodeoxycholic acid
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ursodeoxycholic acid — During 2 years :
  * between 40 and 50 kg : 500 mg/day
  * between 51 and 75 kg : 750 mg/day
  * between 76 and 100 kg : 1000 mg/day
  Other Names: Delursan
  Arms: 1
Drug: Placebo — During 2 years :
  * between 40 and 50 kg : 2 tabs/day
  * between 51 and 75 kg : 3 tabs/day
  * between 76 and 100 kg : 4 tabs/day
  Arms: 2

SUMMARY:
Malignant transformation of adenomas of the duodenum is now the leading cause of death in familial adenomatous polyposis (FAP) patients who had a restorative proctocolectomy. Ursodeoxycholic acid (UDCA) modifies the biliary acid profile and could reduce the severity of duodenal adenomas and prevent such transformation.

DETAILED DESCRIPTION:
We designed a randomized double blinded study to evaluate the efficiency of UDCA in the treatment of duodenal adenomas. One hundred patients are planned to be included. Fifty will receive UDCA and fifty a placebo. Three duodenoscopies are planned: one before inclusion, one at the end of the first year of follow-up and one after two years of follow-up at the end of the protocol. These duodenoscopies are associated to endoscopies of the ileal reservoir performed at the time of restorative proctocolectomy and are recorded numerically. Severity of the duodenal adenomas are evaluated according to the SPIGELMAN score. Patients are seen every 6 months. Before each endoscopy, blood samples are collected for biliary acid profile analysis. Moreover, during endoscopies, duodenal fluid and ileal fluid are collected for biliary acid profile analysis, also.

At the end of the follow-up of the last patients included (nov 2008), biliary acid profile analysis will be performed and statistical analysis of the results will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 18 and 65 years of age
* Weight less than or equal to 100 kg
* Restorative proctocolectomy
* Activated protein C (APC) mutation identified or more than 100 polyps on the colectomy specimen
* SPIGELMAN score of duodenal adenoma greater than or equal to 1
* Efficient contraceptive treatment for pre-menopausal women
* Cooperative patient
* Signed consent
* Social security insurance

Exclusion Criteria:

* SPIGELMAN score of duodenal adenoma equal to 4 with severe dysplasia
* Hepatic disease
* Intermesenteric desmoid tumour
* Any severe disease
* Daily use during the last 3 months of:

  * aspirin;
  * non-steroid anti-inflammatory drugs;
  * tamoxifen;
  * cholestyramine.
* Pregnancy
* Breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2004-10; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
SPIGELMAN severity score of duodenal lesion after 2 years of follow-up | Baseline, 1 and 2 years

SECONDARY OUTCOMES:
Cellular proliferation (Ki 67 and PCNA) | At the baseline, 1 and 2 years
Biliary acid profile | At the baseline, 1 and 2 years
Compliance to the treatment | Every 6 months during 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yann RA Parc, M.D., Ph.D., Principal Investigator — Department of Digestive Surgery, Saint-Antoine Hospital, Hospital of Paris (AP/HP), Pierre et Marie Curie University, 184 rue du Faubourg Saint-Antoine, 75012 Paris, France
Locations (1):
- Saint-Antoine Hospital, Paris, France

REFERENCES:
- [Background] Spigelman AD, Williams CB, Talbot IC, Domizio P, Phillips RK. Upper gastrointestinal cancer in patients with familial adenomatous polyposis. Lancet. 1989 Sep 30;2(8666):783-5. doi: 10.1016/s0140-6736(89)90840-4. PMID 2571019
- [Background] Nugent KP, Farmer KC, Spigelman AD, Williams CB, Phillips RK. Randomized controlled trial of the effect of sulindac on duodenal and rectal polyposis and cell proliferation in patients with familial adenomatous polyposis. Br J Surg. 1993 Dec;80(12):1618-9. doi: 10.1002/bjs.1800801244. PMID 8298943
- [Background] Jarvinen HJ, Nyberg M, Peltokallio P. Biliary involvement in familial adenomatosis coli. Dis Colon Rectum. 1983 Aug;26(8):525-8. doi: 10.1007/BF02563746. PMID 6872780
- [Background] Spigelman AD, Owen RW, Hill MJ, Phillips RK. Biliary bile acid profiles in familial adenomatous polyposis. Br J Surg. 1991 Mar;78(3):321-5. doi: 10.1002/bjs.1800780318. PMID 1850640
- [Background] Mower HF, Ray RM, Shoff R, Stemmermann GN, Nomura A, Glober GA, Kamiyama S, Shimada A, Yamakawa H. Fecal bile acids in two Japanese populations with different colon cancer risks. Cancer Res. 1979 Feb;39(2 Pt 1):328-31. PMID 761204
- [Background] Hill MJ, Drasar BS, Williams RE, Meade TW, Cox AG, Simpson JE, Morson BC. Faecal bile-acids and clostridia in patients with cancer of the large bowel. Lancet. 1975 Mar 8;1(7906):535-9. doi: 10.1016/s0140-6736(75)91556-1. PMID 47015
- [Background] Tanida N, Hikasa Y, Shimoyama T, Setchell KD. Comparison of faecal bile acid profiles between patients with adenomatous polyps of the large bowel and healthy subjects in Japan. Gut. 1984 Aug;25(8):824-32. doi: 10.1136/gut.25.8.824. PMID 6745720
- [Background] van der Werf SD, Nagengast FM, van Berge Henegouwen GP, Huijbregts AW, van Tongeren JH. Colonic absorption of secondary bile-acids in patients with adenomatous polyps and in matched controls. Lancet. 1982 Apr 3;1(8275):759-62. doi: 10.1016/s0140-6736(82)91810-4. No abstract available. PMID 6121223
- [Background] Wilpart M, Mainguet P, Maskens A, Roberfroid M. Structure-activity relationship amongst biliary acids showing comutagenic activity towards 1,2-dimethylhydrazine. Carcinogenesis. 1983 Oct;4(10):1239-41. doi: 10.1093/carcin/4.10.1239. PMID 6616753
- [Background] Earnest DL, Holubec H, Wali RK, Jolley CS, Bissonette M, Bhattacharyya AK, Roy H, Khare S, Brasitus TA. Chemoprevention of azoxymethane-induced colonic carcinogenesis by supplemental dietary ursodeoxycholic acid. Cancer Res. 1994 Oct 1;54(19):5071-4. PMID 7923119
- [Background] Serfaty L, De Leusse A, Rosmorduc O, Desaint B, Flejou JF, Chazouilleres O, Poupon RE, Poupon R. Ursodeoxycholic acid therapy and the risk of colorectal adenoma in patients with primary biliary cirrhosis: an observational study. Hepatology. 2003 Jul;38(1):203-9. doi: 10.1053/jhep.2003.50311. PMID 12830003
- [Background] Parc Y, Piquard A, Dozois RR, Parc R, Tiret E. Long-term outcome of familial adenomatous polyposis patients after restorative coloproctectomy. Ann Surg. 2004 Mar;239(3):378-82. doi: 10.1097/01.sla.0000114216.90947.f6. PMID 15075655
- [Derived] Parc Y, Desaint B, Flejou JF, Lefevre JH, Serfaty L, Vienne A, Kotti S, Simon T, Tiret E. The effect of ursodesoxycholic acid on duodenal adenomas in familial adenomatous polyposis: a prospective randomized placebo-control trial. Colorectal Dis. 2012 Jul;14(7):854-60. doi: 10.1111/j.1463-1318.2011.02816.x. PMID 21899713